CLINICAL TRIAL: NCT02848248
Title: A Phase 1 Study of SGN-CD123A in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: A Safety Study of SGN-CD123A in Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN123-001
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Antibody-Drug Conjugate; CD123 Antigen; Drug Therapy; AML; Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGN-CD123A (Experimental): SGN-CD123A every 3 weeks
  Interventions: Drug: SGN-CD123A

INTERVENTIONS:
Drug: SGN-CD123A — Intravenous infusion in 3-week cycles

SUMMARY:
The study will examine the safety profile of SGN-CD123A. The study will test increasing doses of SGN-CD123A given every 3 weeks to patients.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, and preliminary estimate of antitumor activity of SGN-CD123A. The study will be conducted in 2 parts:

1. Part A is the dose-escalation portion of the trial, designed to identify the maximum tolerated dose (MTD) of SGN-CD123A
2. Part B is the dose-expansion portion of the trial, designed to evaluate SGN-CD123A in patients with differing CD123 expression levels

Dose-escalation in Part A will be conducted using a 3+3 study design. Patients with CD123-detectable AML will be enrolled in cohorts at escalating doses of study drug and will receive up to 2 induction cycles of SGN-CD123A treatment at an assigned dose level in 3-week cycles.

After completion of dose-escalation, patients will be enrolled in Part B of the study. Patients enrolled in Part B will receive up to 2 induction cycles of SGN-CD123A treatment at a dose level and frequency determined by results in Part A.

For both Part A and Part B, a third induction cycle may be permitted with the approval of the study medical monitor. If a patient achieves a complete remission or complete remission with incomplete hematologic recovery, optional post-remission cycles of SGN-CD123A may be administered.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory acute myeloid leukemia following at least 2 but no more than 3 prior regimens
* Patients may be eligible after only 1 previous regimen if in a high risk category
* Adequate baseline renal and hepatic function
* Eastern Cooperative Oncology Group Status of 0 or 1
* CD123-detectable leukemia

Exclusion Criteria:

* Cerebral/meningeal disease related to underlying malignancy
* Promyelocytic leukemia
* History of clinically significant pulmonary fibrosis or documented diffusing capacity of the lung for carbon monoxide <50% predicted
* Prior hematopoietic stem cell transplant
* Antileukemia or experimental treatment within 4 weeks of study drug (other than hydroxyurea or 6-mercaptopurine)
* Cardio or cerebral vascular event within 6 months

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of adverse events | Through 1 month following last dose, or end-of-treatment visit whichever is later
Type, incidence, and severity of laboratory abnormalities | Through 1 month following last dose, or end-of-treatment visit whichever is later
Incidence of dose-limiting toxicity | First cycle of treatment, 3 weeks

SECONDARY OUTCOMES:
Blood concentrations of SGN-CD123A, total antibodies, and metabolites | Through 1 month following last dose, or end-of-treatment visit whichever is later
Incidence of antitherapeutic antibodies | Through 1 month following last dose, or end-of-treatment visit whichever is later
Rate of remission | Through 1 month following last dose, or end-of-treatment visit whichever is later
Duration of complete remission | Up to approximately 1 year
Leukemia-free survival | Up to approximately 1 year
Overall survival | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Phoenix Ho, MD, Study Director — Seagen Inc.
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Hospital / University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hudson Valley Hematology and Oncology Associates/New York Medical College, Hawthorne, New York
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li F, Sutherland MK, Yu C, Walter RB, Westendorf L, Valliere-Douglass J, Pan L, Cronkite A, Sussman D, Klussman K, Ulrich M, Anderson ME, Stone IJ, Zeng W, Jonas M, Lewis TS, Goswami M, Wang SA, Senter PD, Law CL, Feldman EJ, Benjamin DR. Characterization of SGN-CD123A, A Potent CD123-Directed Antibody-Drug Conjugate for Acute Myeloid Leukemia. Mol Cancer Ther. 2018 Feb;17(2):554-564. doi: 10.1158/1535-7163.MCT-17-0742. Epub 2017 Nov 15. PMID 29142066